CLINICAL TRIAL: NCT02285621
Title: Validation of a New Generation of Optimized Orthoses for Personalized Treatment of Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Hubert Labelle, MD, Orthopedist, researcher, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR_259812; 259812 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2014-09-05; First posted 2014-11-07 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Scoliosis; Adolescent Idiopathic Scoliosis (AIS)
Keywords: Scoliosis; Spine deformity; Brace; 3D
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimized brace (Experimental): Test group: Patient will receive optimized brace (3D computer assisted design of the brace)
  Interventions: Other: Optimized brace versus conventional Boston brace
- Standard brace (Active Comparator): Control goup: Patient will receive the Boston Thoracolumbosacral orthosis (TLSO) (conventional design method)
  Interventions: Other: Optimized brace versus conventional Boston brace

INTERVENTIONS:
Other: Optimized brace versus conventional Boston brace — Surface topography using Inspeck cameras allows production of a 3D reconstruction of the patient's trunk, this reconstruction will help to produce the optimized brace. Radiographic and patient-reported data will be gathered and analyzed to observe changes between time points. All radiographs will be taken with an EOS imaging system to allow 3D reconstructions. The SRS-22r will be collected at all clinical visits. Study questions will be aligned as much as possible with other prospective scoliosis protocols so as to minimize patient and surgeon response burden. The study protocol requires no additional visits or radiographs beyond standard of care. Ibuttons are installed in each brace and used to measure the compliance of the patient.

SUMMARY:
Adolescent Idiopathic scoliosis affects 3-4% of the Canadian population, of which about 10% will need a brace treatment during pubertal growth spurt. The design is made relatively corsets empirically, hence the relative efficiency of this treatment. Our team has developed innovative methods for design, optimization and computer aided manufacturing-based numerical simulation models customized to each patient, and a system of evaluation and adjustment of corsets. In this project, the investigators will evaluate the effectiveness of this platform customized treatment and demonstrate its clinical application

ELIGIBILITY:
Inclusion Criteria:

* 10 years or older
* AIS diagnosis
* Risser 0-2
* Primary curve angles 20 degrees - 40 degrees
* If female, either premenarchal or less than 18 months postmenarchal.

Exclusion Criteria:

* Patients with a pre-existing cardiovascular condition
* Patients with symptom of a neurological disorder
* Patients with any other disorder of the musculoskeletal system affecting the lower limbs,

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Change in Cobb angle | Baseline, 6 months, 1 year
  Radiographics will be gathered and analyzed to observe changes between time points. All radiographs will be taken with an low-dose biplane radiographic system (EOS) to allow 3D reconstructions.

SECONDARY OUTCOMES:
Change in Scoliosis Research Society questionnaire (SRS-22r) scores | Baseline, 6 months, 1 year
  The SRS-22r questionnaire is available from SRS.org. It is a self-reported tools assessing self-image, function, pain, mental health with 5 questions each and satisfaction with care with 2 questions. A total score is also available based on all 22 questions.
Change in surface topography | Baseline, 6 months, 1 year
  Four optical scanners are used to capture full trunk images. Subjects are positioned in a standard frame, and reference points marked. Parameters quantifying the external back surface deformity are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Labelle, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Cobetto N, Aubin CE, Parent S, Barchi S, Turgeon I, Labelle H. 3D correction of AIS in braces designed using CAD/CAM and FEM: a randomized controlled trial. Scoliosis Spinal Disord. 2017 Jul 23;12:24. doi: 10.1186/s13013-017-0128-9. eCollection 2017. PMID 28770254
- [Derived] Cobetto N, Aubin CE, Parent S, Clin J, Barchi S, Turgeon I, Labelle H. Effectiveness of braces designed using computer-aided design and manufacturing (CAD/CAM) and finite element simulation compared to CAD/CAM only for the conservative treatment of adolescent idiopathic scoliosis: a prospective randomized controlled trial. Eur Spine J. 2016 Oct;25(10):3056-3064. doi: 10.1007/s00586-016-4434-3. Epub 2016 Feb 9. PMID 26861663